CLINICAL TRIAL: NCT03736785
Title: A Phase 2, Randomized, Open-Label Trial to Evaluate the Safety and Efficacy of LY3209590 in Study Participants With Type 2 Diabetes Mellitus Previously Treated With Basal Insulin
Brief Title: A Study of LY3209590 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17059; I8H-MC-BDCM (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3209590 Algorithm 1 (Experimental): Participants received loading dose followed by weekly dose of LY3209590 based on the prior randomization basal insulin dose for a period of 32 weeks by subcutaneous (SC) injection. Dose titration was done to maintain fasting blood glucose of <140 milligram per deciliter (mg/dL).
  Interventions: Drug: LY3209590
- LY3209590 Algorithm 2 (Experimental): Participants received loading dose followed by weekly dose of LY3209590 based on the prior randomization basal insulin dose for a period of 32 weeks by subcutaneous injection. Dose titration was done to maintain fasting blood glucose of <120 mg/dL.
  Interventions: Drug: LY3209590
- Insulin Degludec (Active Comparator): Participants received same dose of Degludec as the total basal insulin dose already administered prior to randomization. Dose was titrated to maintain fasting blood glucose of ≤100 mg/dL to achieve glycemic goal of HbA1C <7%.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590 Algorithm 1; LY3209590 Algorithm 2
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Degludec

SUMMARY:
The reason for this study is to see if the study drug LY3209590 is safe and effective in participants with type 2 diabetes that have already been treated with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus according to the World Health Organization (WHO) criteria treated with basal insulin and up to 3 of the following oral antihyperglycemic medication (OAM):

  * dipeptidyl peptidase-4 (DPP-4) inhibitors
  * sodium-glucose cotransporter (SGLT-2) inhibitors
  * biguanides
  * alpha-glucosidase inhibitors
  * sulfonlyureas
* HbA1c value of 6.5% to 10%, inclusive
* Body mass index (BMI) between 20 and 45 kilograms per meter squared (kg/m2), inclusive

Exclusion Criteria:

* Type 1 diabetes mellitus or latent autoimmune diabetes
* Any episodes of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening
* Any of the following cardiovascular (CV) conditions: acute myocardial infarction, New York Heart Association Class III or IV heart failure, or cerebrovascular accident (stroke)
* Acute or chronic hepatitis, or obvious clinical signs or symptoms of any other liver disease
* Estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 m2
* Active or untreated malignancy
* Chronic (>14 days) systemic glucocorticoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- United States (36):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Arkansas Clinical Research, Little Rock, Arkansas
  - John Muir Physician Network Clinical Research Center, Concord, California
  - AMCR Institute INC, Escondido, California
  - Valley Endocrine, Fresno, Fresno, California
  - Marin Endocrine Associates, Greenbrae, California
  - National Research Institute, Huntington Park, California
  - First Valley Medical Group, Lancaster, California
  - National Research Institute, Los Angeles, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Metabolic Research Institute Inc., West Palm Beach, Florida
  - East West Medical Institute, Honolulu, Hawaii
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Iderc, P.L.C., West Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Metrolina Internal Medicine, P.A., Charlotte, North Carolina
  - Intend Research, Norman, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians - Jacob Murphy Lane, Uniontown, Pennsylvania
  - Internal Medicine Associates of Anderson, Anderson, South Carolina
  - The Research Center of the Upstate, Mauldin, South Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Confluence Health Clinical Research Department, Wenatchee, Washington
- Mexico (2):
  - Hospital Universitario UANL, Monterrey, Nuevo León
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
- Puerto Rico (5):
  - Advanced Clinical Research, LLC, Bayamón, PR
  - Manati Center for Clinical Research Inc, Manatí, PR
  - GCM Medical Group PSC, San Juan, PR
  - Martha Gomez Cuellar M.D., San Juan, PR
  - Centro de Endocrinologia del Este, Yabucoa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Frias J, Chien J, Zhang Q, Chigutsa E, Landschulz W, Syring K, Wullenweber P, Haupt A, Kazda C. Safety and efficacy of once-weekly basal insulin Fc in people with type 2 diabetes previously treated with basal insulin: a multicentre, open-label, randomised, phase 2 study. Lancet Diabetes Endocrinol. 2023 Mar;11(3):158-168. doi: 10.1016/S2213-8587(22)00388-6. Epub 2023 Feb 6. PMID 36758572
- See also: A Study of LY3209590 in Participants With Type 2 Diabetes Mellitus — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/BDCM

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3209590 Algorithm 1: Participants received loading dose followed by weekly dose of LY3209590 based on the prior randomization basal insulin dose for a period of 32 weeks by subcutaneous (SC) injection. Dose titration was done to maintain fasting blood glucose of <140 mg/dL.
Period: Overall Study
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Started | 135 | 132 | 132
Completed | 118 | 115 | 118
Not Completed | 17 | 17 | 14
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Death | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Non compliance with study drug | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 4 | 3
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Unknown/Missing data | 3 | 2 | 1
Not completed — Withdrawal by Subject | 9 | 6 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY3209590 Algorithm 1: Participants received loading dose followed by weekly dose of LY3209590 based on the prior randomization basal insulin dose for a period of 32 weeks by subcutaneous (SC) injection. Dose titration was done to maintain fasting blood glucose of <140 milligram mg.dL
- Total: Total of all reporting groups
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec | Total
Number analyzed (Participants) | 135 | 132 | 132 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.9) | 59.6 (11.3) | 60.8 (10.0) | 60.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 65 | 202
  Male | 68 | 62 | 67 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 78 | 73 | 218
  Not Hispanic or Latino | 68 | 54 | 59 | 181
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 18 | 19 | 53
  Asian | 4 | 5 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 16 | 10 | 10 | 36
  White | 97 | 97 | 94 | 288
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 18 | 16 | 15 | 49
  United States | 96 | 97 | 96 | 289
  Mexico | 21 | 19 | 21 | 61
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: HbA1C percentage (%)] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  HbA1C percentage (%) | 8.20 (0.87) | 8.03 (0.89) | 8.13 (0.88) | 8.12 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: HbA1c is the glycosylated fraction of haemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Change from baseline in HbA1c was analysed by mixed model repeated measures (MMRM) including fixed effects of treatment, stratification factors (country, BMI group [> 30 or ≤ 30], sulfonylureas use at study entry), visit and treatment by visit interaction and baseline HbA1c as the covariate.
Time Frame: Baseline, Week 32
Population: The data after using rescue medication or stopping study medication were censored. Participants with non-missing baseline value and at least one post baseline value of response were included.
Measure: Least Squares Mean (Standard Error); unit: HbA1C %
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Number analyzed (Participants) | 130 | 125 | 124
HbA1C % | -0.58 (0.083) | -0.57 (0.085) | -0.66 (0.084)
Statistical Analysis 1: Comparison: LY3209590 Algorithm 1; Test type: Equivalence — Equivalence margin is zero; p < 0.001, Mixed Models Analysis — P-value reported is within group comparison between Week 32 and baseline
Statistical Analysis 2: Comparison: LY3209590 Algorithm 2; Test type: Equivalence — Equivalence margin is zero; p < 0.001, Mixed Models Analysis — P-value reported is within group comparison between Week 32 and baseline
Statistical Analysis 3: Comparison: Insulin Degludec; Test type: Equivalence — Equivalence margin is zero; p < 0.001, Mixed Models Analysis — P-value reported is within group comparison between Week 32 and baseline

2. Secondary Outcome: Change From Baseline in HbA1c Compared to Insulin Degludec
Description: HbA1c is the glycosylated fraction of haemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Change from baseline in HbA1c was analysed by MMRM including fixed effects of treatment, stratification factors (country, BMI group [> 30 or ≤ 30], sulfonylureas use at study entry), visit and treatment by visit interaction, and baseline HbA1c as the covariate.
Time Frame: Baseline, Week 32
Population: The data after using rescue medication or stopping study medication were excluded. Participants with non-missing baseline value and at least one post baseline value of response were included.
Measure: Least Squares Mean (Standard Error); unit: HbA1C %
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Number analyzed (Participants) | 130 | 125 | 124
HbA1C % | -0.58 (0.083) | -0.57 (0.085) | -0.66 (0.084)
Statistical Analysis 1: Comparison: LY3209590 Algorithm 1 vs Insulin Degludec; Test type: Non-Inferiority — Non-inferiority margin is 0.4%; Mixed Models Analysis; LSMean Difference = 0.08, 90% CI 2-sided [-0.11 to 0.28]
Statistical Analysis 2: Comparison: LY3209590 Algorithm 2 vs Insulin Degludec; Test type: Non-Inferiority — Non-inferiority margin is 0.4%; Mixed Models Analysis; LSMean Difference = 0.09, 90% CI 2-sided [-0.10 to 0.29]

3. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Change from baseline in fasting glucose was analysed by MMRM including fixed effects of treatment, stratification factors (country, BMI group [> 30 or ≤ 30], sulfonylureas use at study entry, HbA1c strata [<8.5% or ≥8.5%]), visit and treatment by visit interaction, and baseline fasting glucose as the covariate.
Time Frame: Baseline, Week 32
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milligram per deicliter (mg/dL)
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Number analyzed (Participants) | 130 | 125 | 124
Milligram per deicliter (mg/dL) | -13.1 (4.01) | -18.6 (4.14) | -31.5 (4.03)

4. Secondary Outcome: Change From Baseline in Insulin Dose (LY3209590)
Description: The baseline for both LY3209590 arms was the first regular weekly dose at Week 1.
Time Frame: Week 1, Week 32
Population: Participants with non-missing value at the specified timepoint were included.The data after using rescue medication or stopping study medication were excluded.
Measure: Mean (Standard Deviation); unit: Milligrams (mg)
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2
Number analyzed (Participants) | 118 | 115
Milligrams (mg) | 0.12 (4.86) | 0.60 (3.75)

5. Secondary Outcome: Change From Baseline in Insulin Dose (Insulin Degludec)
Description: Change from Baseline in Insulin Dose for Insulin Degludec arm was reported.
Time Frame: Baseline, Week 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Insulin Degludec
Number analyzed (Participants) | 111
International Units (IU) | 16.40 (26.06)

6. Secondary Outcome: Rate of Total Documented Symptomatic Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with glucose ≤54 mg/dL (3.0 millimole per liter (mmol/L)). Relative Rate was calculated based on Group Mean. Group Mean was estimated by first taking the inverse link function on individual patient covariates, then averaging over all participants.
Time Frame: Baseline through week 32
Population: All randomized study participants who received at least one dose of study medication and had evaluable hypoglycaemic data.
Measure: Mean (Standard Error); unit: Events per participant per year
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Number analyzed (Participants) | 135 | 131 | 132
Events per participant per year | 0.73 (0.119) | 1.22 (0.378) | 1.56 (0.375)

7. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was analysed by MMRM including fixed effects of treatment, visit and treatment by visit interaction, and baseline body weight as the covariate.
Time Frame: Baseline, Week 32
Population: All randomized participants who received at least one dose of study medication and with non-missing baseline value and at least one post baseline value of response were included.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
Number analyzed (Participants) | 135 | 130 | 129
Kilogram (kg) | 1.0 (0.33) | 1.0 (0.33) | 2.0 (0.33)

8. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3209590
Description: PK: AUC of LY3209590 was reported for LY3209590 Algorithm 1 and LY3209590 Algorithm 2 arms. AUC was calculated for individual participants using the participant's Week 32 LY3209590 dose amount and the participant's estimated clearance value.
Time Frame: Week 32
Population: All randomized participants who received at least one dose of LY3209590 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole * hour per Liter (nmol * hr/L)
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2
Number analyzed (Participants) | 119 | 112
Nanomole * hour per Liter (nmol * hr/L) | 5360 (67) | 5430 (60)

ADVERSE EVENTS:
Time Frame: Up to 37 weeks
Description: All randomized participants.
Arm/Group | LY3209590 Algorithm 1 | LY3209590 Algorithm 2 | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 1/135 | 0/132 | 1/132
Serious Adverse Events (participants affected / at risk) | 7/135 | 8/132 | 10/132
Other Adverse Events (participants affected / at risk) | 17/135 | 29/132 | 13/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3209590 Algorithm 1 (N=135) | LY3209590 Algorithm 2 (N=132) | Insulin Degludec (N=132)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3209590 Algorithm 1 (N=135) | LY3209590 Algorithm 2 (N=132) | Insulin Degludec (N=132)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 8 (9) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 14 (14) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT03736785/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03736785/SAP_001.pdf